CLINICAL TRIAL: NCT00908960
Title: A Randomized Controlled Trial of Enoxaparin Thromboprophylaxis in Cancer Patients With Elevated Tissue Factor Bearing Microparticles
Brief Title: Enoxaparin Thromboprophylaxis in Cancer Patients With Elevated Tissue Factor Bearing Microparticles
Acronym: MicroTEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); North Shore Medical Center (Other); University of Southern California (Other); VA Boston Healthcare System (U.S. Federal Agency); Sanofi (Industry)
Responsible Party: Principal Investigator, Jeffrey Zwicker, MD, Attending Physician, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-378
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Advanced Pancreatic, Colon, Lung, Gastric and Ovarian Cancer
Keywords: enoxaparin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High TFMP: Enoxaparin (Experimental): Patients received enoxaparin 40 mg subcutaneously once daily for 2 months (60 days).Only patients with high TFMP status at baseline were randomized to treatment or observation.
  Interventions: Drug: Enoxaparin
- High TFMP: Observation (No Intervention): Patients undergo observation until evaluation with a lower extremity ultrasound at 2 months (day 60). Only patients with high TFMP status at baseline were randomized to treatment or observation.
- Low TFMP: Observation (No Intervention): Patients undergo observation until evaluation with a lower extremity ultrasound at 2 months (day 60). Patients with low TFMP status at baseline were directly assigned to observation.

INTERVENTIONS:
Drug: Enoxaparin
  Other Names: Lovenox
  Arms: High TFMP: Enoxaparin

SUMMARY:
Research studies have shown a strong association between cancer and blood clots in the veins (also known as deep vein thrombosis). These blood clots can flow to the lungs (pulmonary embolism) which in severe cases may be life threatening. The purpose of this research study is to see if enoxaparin is effective in preventing blood clots in the veins in participants who have cancer of the pancreas, colorectal, non-small cell lung, ovary, or gastric and also have high levels of tissue factor bearing microparticles in their blood (TFMP). TFMP are small particles that are generated from different types of blood cells in the body. In people who have cancer, TFMP are thought to be generated from cancer cells and may represent a risk factor for deep vein thrombosis. Enoxaparin has been used to prevent formation of blood clots in patients after abdominal or orthopedic surgery and in patients who suffer from a severe medical illness. Based on these studies, we are investigating to see if it prevents thrombosis in people with certain types of cancer.

DETAILED DESCRIPTION:
The study was a randomized phase II trial to evaluate the cumulative incidence of VTE in cancer outpatients. At baseline, measurement of tissue factor-bearing microparticles (TFMP) was performed by impedance-based flow cytometry based on established methods. (Zwicker et al, 2009) Patients were classified as having high or low TFMP levels based on a reference repository of plasmas from sixty cancer patients. The top tercile of tissue factor-bearing microparticle concentrations from the reference specimens (3.5 x 104 microparticles/µl) was considered a cutoff for "high" and corresponds with previously described "detectable" levels. Patients with high levels were randomized (2:1) to enoxaparin 40 mg subcutaneously once daily or observation. Randomization was stratified based on cancer diagnosis. Low TFMP patients were observed without anticoagulation. Both the treating physicians and patients were blinded to microparticle status in the observation arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy that is metastatic or unresectable and for which standard curative therapies do not exist. Eligible malignancies include:

  * Adenocarcinoma of the pancreas (locally advanced or metastatic)
  * Colorectal (stage IV)
  * Non-small cell lung (unresectable stage III or IV)
  * Relapsed ovarian or stage IV
  * Surgically unresectable or metastatic gastric adenocarcinoma
* First or second line therapy (within 4 weeks of initiating therapy).
* Minimum age 18 years
* Life expectancy of greater than 6 months
* ECOG Performance Status 0, 1, or 2 (Karnofsky 60% or greater).
* Participants must have normal organ and marrow function as outlined in the protocol.

Exclusion Criteria:

* Participants may not be receiving any other study agents.
* Known brain metastases should be excluded from this clinical trial because of their poor prognosis and higher potential for intracranial hemorrhage.
* Prior history of documented venous thromboembolic event or pulmonary embolism within the last 5 years years (excluding central line associated events whereby patients completed anticoagulation > 3 months previously)
* Active bleeding or high risk for bleeding (e.g. known acute gastrointestinal ulcer)
* Any history of significant hemorrhage (requiring hospitalization or transfusion) outside of a surgical setting within the last 5 years
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enoxaparin or heparin.
* History of heparin-induced thrombocytopenia
* Presence of coagulopathy (PT or PTT> 1.5 x upper limit of normal)
* Familial bleeding diathesis
* Known diagnosis of disseminated intravascular coagulation
* Currently receiving anticoagulant therapy
* Current use of aspirin (>81mg daily), Clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox), or regular use of non-steroidal anti-inflammatory agents more than twice weekly. Maximum dose of ibuprofen is 400mg no more than twice per week.
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zwicker, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- United States (5):
  - University of Southern California-Keck School of Medicine, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - VA Boston Healthcare System, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts

REFERENCES:
- [Result] Zwicker JI, Liebman HA, Bauer KA, Caughey T, Campigotto F, Rosovsky R, Mantha S, Kessler CM, Eneman J, Raghavan V, Lenz HJ, Bullock A, Buchbinder E, Neuberg D, Furie B. Prediction and prevention of thromboembolic events with enoxaparin in cancer patients with elevated tissue factor-bearing microparticles: a randomized-controlled phase II trial (the Microtec study). Br J Haematol. 2013 Feb;160(4):530-7. doi: 10.1111/bjh.12163. Epub 2012 Dec 13. PMID 23240761
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539

RESULTS

PARTICIPANT FLOW:
Groups:
- High TFMP: Enoxaparin: Patients received enoxaparin 40 mg subcutaneously once daily for 2 months (60 days). Only patients with high TFMP status at baseline were randomized to treatment or observation.
- High TFMP: Observation: Patients undergo observation until evaluation with lower extremity ultrasound at 2 months (day 60). Only patients with high TFMP status at baseline were randomized to treatment or observation.
- Low TFMP: Observation: Patients undergo observation until evaluation with lower extremity ultrasound at 2 months (day 60). Patients with low TFMP status at baseline were directly assigned to observation.
Period: Overall Study
Arm/Group | High TFMP: Enoxaparin | High TFMP: Observation | Low TFMP: Observation
Started | 24 | 12 | 34
Evaluable | 23 | 11 | 32
Completed | 23 | 11 | 32
Not Completed | 1 | 1 | 2
Not completed — Presence VTE dx or Absent VTE eval | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all evaluable patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | High TFMP: Enoxaparin | High TFMP: Observation | Low TFMP: Observation | Total
Number analyzed (Participants) | 23 | 11 | 32 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 19 | 33
  >=65 years | 13 | 7 | 13 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.5) | 63.4 (15.0) | 63.3 (11.7) | 64.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 13 | 28
  Male | 14 | 5 | 19 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 11 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: 2-Month Cumulative Incidence of VTE
Description: 2-month cumulative incidence of venous thromboembolism (VTE) is the probability of experiencing within 2 months of study entry the following events: any symptomatic proximal or distal lower extremity deep vein thrombosis, symptomatic pulmonary embolism or fatal pulmonary embolism diagnosed by autopsy, or asymptomatic proximal deep vein thrombosis diagnosed by screening compression ultrasound.
Time Frame: Assessment with lower extremity ultrasound occured at day 60/ month 2
Population: The analysis dataset is comprised of all evaluable patients.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | High TFMP: Enoxaparin | High TFMP: Observation | Low TFMP: Observation
Number analyzed (Participants) | 23 | 11 | 32
percent probability | 5.6 [0 to 16.6] | 27.2 [0 to 55.1] | 7.2 [0 to 17.1]
Statistical Analysis 1: Comparison: High TFMP: Enoxaparin vs High TFMP: Observation; Test type: Superiority or Other; p = 0.06, Fine and Gray regression; Hazard Ratio (HR) = 6.7, 95% CI 2-sided [1.03 to 43.17]

2. Secondary Outcome: Incidence of Major Hemorrhage Events
Description: Incidence is the number of patients experiencing at least one major hemorrhage events as defined according to International Society on Thrombosis and Haemostasis (ISTH) guidelines. (Schulman and Kearon 2005)
Time Frame: Assessed during the 60 day therapy
Population: The analysis dataset is comprised of evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | High TFMP: Enoxaparin | High TFMP: Observation | Low TFMP: Observation
Number analyzed (Participants) | 23 | 11 | 32
Participants | 0 | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive and estimated using Kaplan-Meier (KM) methods.
Time Frame: Assessed up to approximately 30 months
Population: The analysis dataset is comprised of all evaluable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | High TFMP: Enoxaparin | High TFMP: Observation | Low TFMP: Observation
Number analyzed (Participants) | 23 | 11 | 32
months | 17.8 [5.2 to 30] | 11.8 [5.4 to 18.2] | 17.3 [10.3 to 24.3]

ADVERSE EVENTS:
Time Frame: Assessed during the 60 day therapy
Arm/Group | High TFMP: Enoxaparin | High TFMP: Observation | Low TFMP: Observation
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/11 | 0/32
Other Adverse Events (participants affected / at risk) | 6/23 | 2/11 | 7/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High TFMP: Enoxaparin (N=23) | High TFMP: Observation (N=11) | Low TFMP: Observation (N=32)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) — A subject with lung cancer on the observation arm experienced shortness of breath while on trial. Another study subject with pancreatic cancer on the observation arm died following rapidly progressive shortness of breath and hypoxia at nursing home.
Disease progression (Investigations) | 2 (2) | 1 (1) | 3 (3) — These subjects had disease progression: 3 Lung cancer on observation; 1 pancreatic cancer on observation; 1 pancreatic cancer on lovenox and another lung cancer on lovenox.
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — A pancreatic cancer subject on observation arm died following a blood infection.
Platelets (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) — Subject with lung cancer on lovenox and was found with low platelets. Another subject with colon cancer on observation was also found with low platelets.
Alkaline Phosphotase and aspartate aminotransferase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Subject with pancreatic cancer and on lovenox was hospitalized for a decreased urine output, obstructive liver function tests, and ankle edema.
Lymphatics (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Subject with lung cancer and on lovenox was hospitalized with increased swelling and discomfort over left side of neck.
pneumonia and anemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — subject with pancreatic cancer on lovenox arm was hospitalized for pneumonia and anemia.
elevated troponin (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — A pancreatic cancer subject on observation arm with elevated troponin
GI-Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Study subject with pancreatic cancer on the observation arm died following an gastrointestinal bleed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No